CLINICAL TRIAL: NCT03059238
Title: Study of Parecoxib Versus Celecoxib Versus Oxycodone on Perioperative Pain Control of Transcatheter Chemoembolization Procedure for Patients With Hepatocelullar Carcinoma
Brief Title: Parecoxib Versus Celecoxib Versus Oxycodone in Pain Control for Transcatheter Chemoembolization Procedure
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Ming Zhao, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016-FXY-099
Record Dates: First submitted 2017-02-10; First posted 2017-02-23 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Liver Cancer; Pain Postoperative
Keywords: Pain control; TACE; Opioids; NSAIDs
MeSH Terms: conditions — Liver Neoplasms; Pain, Postoperative; Agnosia | interventions — Celecoxib; parecoxib

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Celecoxib group (Experimental): Celecoxib 200mg oral capsule, 200 mg, orally one hour before TACE and once every 12 hours for 2 days after TACE, with totally 5 times.
  Interventions: Drug: Celecoxib 200mg oral capsule
- Parecoxib group (Experimental): Parecoxib sodium , 40 mg, dissolved in 3 mL 0.9% sodium chloride intravenously one hour before TACE and once every 12 hours for 2 days after TACE, with totally 5 times.
  Interventions: Drug: parecoxib sodium
- Oxycodone group (Experimental): Controlled-release oxycodone, 10 mg, orally one hour before TACE and once every 12 hours for 2 days after TACE, with totally 5 times.
  Interventions: Drug: controlled-release oxycodone

INTERVENTIONS:
Drug: Celecoxib 200mg oral capsule
  Arms: Celecoxib group
Drug: parecoxib sodium
  Arms: Parecoxib group
Drug: controlled-release oxycodone
  Arms: Oxycodone group

SUMMARY:
This phase III, randomized, prospective clinical study, aiming to compare the analgesic effects of celecoxib, parecoxib, and oxycodone in patients with inoperable hepatic carcinoma undergoing TACE procedure in postoperative pain control.

DETAILED DESCRIPTION:
Studies reported that almost 75% of patients with hepatocellular carcinoma undergoing transcatheter arterial chemoembolization (TACE) experienced severe pain (in a three-grade mild, moderate, and severe classification), and 93% of patients required opioid treatment during the first 12 hours after TACE.

Opioids and nonsteroidal anti-inflammatory drugs (NSAIDs) are most commonly used analgesic medications in the control of postoperative surgical pain. Previous studies has indicated that both controlled-release oxycodone, which is an oral semisynthetic opioid µ and κ agonist, and parecoxib sodium, a parenteral COX-2 selective inhibitor, were effective and safe on peri- and post-procedural pain in HCC patients undergoing TACE.

To the investigators's knowledge, no studies have been developed on comparing differences of efficacy and feasibility of analgesics with different action mechanism (opioids vs. NSAIDs) and administration route (oral path vs. injective path) on pain control for patients undergone TACE. In this phase III, randomized, prospective clinical study, the investigators aimed to compare the analgesic effects of celecoxib (oral NSAIDs), parecoxib (injective NSAIDs), and controlled-release oxycodone (oral opioids) in patients with inoperable hepatic carcinoma undergoing TACE procedure in postoperative pain control.

ELIGIBILITY:
Inclusion Criteria:

* Patients included in the study were classified with stage B or C according to the Barcelona Clinic Liver Cancer (BCLC) staging classification.
* Patients were recommended to receive TACE therapy for HCC.

Exclusion Criteria:

* hypersensitive to celecoxib, parecoxib, and oxycodone
* a history of serious allergic reactions to medicines
* stomach ulcers or bleeding in the stomach or gut
* allergic-type reactions such as bronchospasm, cold-like symptoms, polyps in the nose, swelling of the face or hives after taking aspirin or NSAIDs, including other COX-2 inhibitors
* severe liver disease
* inflammatory bowel disease
* heart failure, ischaemic heart disease, peripheral artery disease, or cerebrovascular disease
* women during the last three months of pregnancy or to breast-feeding women
* after coronary surgery

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Pain score | 48 hours
  Self reported pain intensity using the numeric rating scale (NRS) (score of 0-10) after administration of the first dose of study medication.

SECONDARY OUTCOMES:
Adverse events | 48 hours
  Adverse events scores of fever, vomiting, nausea, constipation, dysuria, and hypersomnia were rated according to the National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0.
Trouble sleeping | 48 hours
  Self reported sleep trouble using the numeric rating scale 1-4 (1 = not at all; 2 = a little; 3 = quite a bit; 4 = very much) once every 24 hours after administration of the first dose of study medication.
Fatigue | 48 hours
  Self reported fatigue using the numeric rating scale 1-4 (1 = not at all; 2 = a little; 3 = quite a bit; 4 = very much) once every 24 hours after administration of the first dose of study medication.
Lacked appetite | 48 hours
  Self reported lacked appetite using the numeric rating scale 1-4 (1 = not at all; 2 = a little; 3 = quite a bit; 4 = very much) once every 24 hours after administration of the first dose of study medication.
Spiritual state | 48 hours
  Self reported fatigue using the numeric rating scale 1-4 (1 = Very well; 2 = normal; 3 = poor; 4 = worst) once every 24 hours after administration of the first dose of study medication.

CONTACTS AND LOCATIONS:
Overall Officials: Ming Zhao, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Minimally Invasive Interventional Division, Department of Medical Imaging and Interventional Radiology, Sun Yat-sen University Cancer Center,, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhou B, Wang J, Yan Z, Shi P, Kan Z. Liver cancer: effects, safety, and cost-effectiveness of controlled-release oxycodone for pain control after TACE. Radiology. 2012 Mar;262(3):1014-21. doi: 10.1148/radiol.11110552. PMID 22357901
- [Background] Zhou ZG, Chen JB, Qiu HB, Wang RJ, Chen JC, Xu L, Chen MS, Zhang YJ. Parecoxib prevents complications in hepatocellular carcinoma patients receiving hepatic transarterial chemoembolization: a prospective score-matched cohort study. Oncotarget. 2016 May 10;7(19):27938-45. doi: 10.18632/oncotarget.8560. PMID 27056892
- [Result] Lv N, Kong Y, Mu L, Pan T, Xie Q, Zhao M. Effect of perioperative parecoxib sodium on postoperative pain control for transcatheter arterial chemoembolization for inoperable hepatocellular carcinoma: a prospective randomized trial. Eur Radiol. 2016 Oct;26(10):3492-9. doi: 10.1007/s00330-016-4207-8. Epub 2016 Jan 22. PMID 26801163